CLINICAL TRIAL: NCT04472754
Title: The Biological Basis of Phlegm Dampness Syndrome in Patients With Ischemic Stroke：A Saliva and Urine Proteomics Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Guangzhou Cadre Health Management Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8388
Record Dates: First submitted 2020-05-21; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-05

CONDITIONS: Protein; Disease
Keywords: ischemic stroke; phlegm dampness syndrome; traditional Chinese medicine; proteomic
MeSH Terms: conditions — Disease; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — All the saliva and urine samples will be stored in the biological resource centre of the our research centre after written informed consent obtained from all subjects who voluntarily participated in this clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A(healthy control group): patients who did not have ischemic stroke and whose TCM constitution was dialectically peaceful;
- B: Patients with no ischemic stroke and whose TCM constitution was dialectical with damp phlegm constitution
- C: patients with ischemic stroke diagnosed with phlegm dampness syndrome
- D: patients with ischemic stroke diagnosed as non-phlegm dampness syndrome

SUMMARY:
This study aimed to explorie the biological basis of phlegm-dampness syndrome in patients with ischemic stroke using proteomics research techniques of urine and saliva.

DETAILED DESCRIPTION:
Stroke is the disease with the highest mortality and disability in China, and the annual incidence of ischemic stroke is the highest. Atherosclerosis is the main cause of ischemic stroke. According to the theory of traditional Chinese medicine, the disease is closely related to the physical constitution of the individual. The main body constitution of the population in Lingnan area is phlegm dampness syndrome;Previous large cross-sectional studies have found that 65.3% of patients with ischemic stroke in Lingnan area have phlegm dampness syndrome. However, there is currently no biological evidence related to phlegm-dampness syndrome and ischemic stroke.In recent years, proteomics research technology has developed vigorously. The research samples have developed from blood obtained from minimally invasive to urine and saliva obtained non-invasively. Studies have found that urine proteins associated with AS include type I, type III collagen, 8-isoprostaglandin F2α, and saliva proteins include IL-1β, IL-6, TNF-α, and PGE2.Therefore, this research is dedicated to exploring the biological basis of phlegm-dampness syndrome in patients with ischemic stroke using proteomics research techniques of urine and saliva.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ischemic stroke
2. Aged 35-80-year-old.
3. Agree to participate in clinical research and sign informed consent.

Exclusion Criteria:

1. Clinical diagnosis of cerebral hemorrhage;
2. With severe infection, severe renal dysfunction, and tumor;
3. Clinical diagnosis of acute oral inflammation, oral ulcers, or urinary infections;
4. Clinical diagnosis of systemic lupus erythematosus and rheumatoid arthritis;
5. Pregnant women or lactating mothers

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population are people who diagnosed as ischemic stroke at Guangdong Provincial Hospital of Chinese Medicine The healthy volunteers are definted as people who have no history of cerebrovascular diseases (including cerebral hemorrhage, cerebral infarction, transient ischemic attack, etc.)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Differentially expressed proteins of urine and saliva | 1 day
  Proteomic expression of urine and saliva in each group will be tested use Protein liquid chromatography/mass spectrometry detection.

SECONDARY OUTCOMES:
NIHSS scoes | 1 day
  NIHSS scoring scale for neurological impairment assessment
modified Rankin Scale (mRS) score | 1 day
  mRS score for the degree of dependence
BI index | 1 day
  BI index for living ability assessment